CLINICAL TRIAL: NCT00242216
Title: "PIQD: The Once a Day Protease Inhibitor Regimens." Ritonavir Boosted Atazanavir vs. Ritonavir Boosted Fosamprenavir Used in Combination With Tenofovir and Emtricitabine in HIV-1 Infected Antiretroviral Treatment-Naïve Patients.
Brief Title: "The Once A Day Protease Inhibitor Regimens"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Roberto Arduino, Professor - Internal Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-03-315
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
Keywords: HIV-1 infected people; Antiretroviral treatment-naïve; Atazanavir; Fosamprenavir; ARV Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir; fosamprenavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atazanavir oral once daily (Active Comparator): HIV treatment
  Interventions: Drug: ritonavir-boosted atazanavir
- Fosamprenavir oral once daily (Active Comparator): HIV treatment
  Interventions: Drug: ritonavir-boosted fosamprenavir

INTERVENTIONS:
Drug: ritonavir-boosted atazanavir — 100 mg ritonavir plus 300 mg atazanavir in combination with tenofovir-emtricitabine fixed dose combination given once daily.
  Other Names: Reyataz plus Norvir
  Arms: Atazanavir oral once daily
Drug: ritonavir-boosted fosamprenavir — 100 mg ritonavir plus 1,400 mg fosamprenavir in combination with tenofovir-emtricitabine fixed dose combination given once daily.
  Other Names: Lexiva plus Norvir
  Arms: Fosamprenavir oral once daily

SUMMARY:
Atazanavir (ATV) and fosamprenavir (fAPV) are new protease inhibitors that can be administered once-a-day and boosted with ritonavir (r). Prior studies have demonstrated that both are effective in treatment of ARV-naïve HIV-infected people. This study was designed to demonstrate if a HAART regimen containing ATV/r is not inferior to a HAART regimen containing fAPV/r, in ARV-naïve patients over a 96-week period.

This is a phase IV, single center, randomized, open label, 2-arm clinical trial in ARV therapy-naïve patients with HIV-1 RNA >1,000 copes/mL and CD4 cell count <350 cells/mm3. Patients will be randomized to receive tenofovir and emtricitabine plus either ATV (300mg qd) and ritonavir (100mg qd) or fAPV (1400mg qd) and ritonavir (200mg qd).

DETAILED DESCRIPTION:
Over the past decade, there have been significant advances toward fighting the progression of HIV disease. Current treatment strategies consist of utilization of potent combination antiretroviral therapy to suppress HIV replication below detectable limits limiting the potential for the emergence of resistant viruses, boosting CD4 cell counts and thereby delaying disease progression. Treatment of HIV-1 infection with Highly Active Antiretroviral Therapy (HAART) regimens containing a protease inhibitor (PI) and two nucleoside reverse transcriptase inhibitor (NRTIs) has been shown to prolong survival and decrease disease progression. Despite these potent antiretroviral agents, current available therapies continue to fail in some patients. Poor adherence to complex treatment regimens remains a significant cause of suboptimal viral suppression leading to emerge of resistant virus. Atazanavir and fosamprenavir were recently FDA approved protease inhibitors. The efficacy and safety profile of these two drugs have been established in clinical trials enrolling antiretroviral therapy naïve and protease inhibitor experienced patients. Atazanavir and fosamprenavir are the only protease inhibitors approved for a once a day regimen and this may set a new standard for treatment of antiretroviral therapy naïve HIV infected patients. Adherence to the medicines, a key component of treatment success, could be significantly improved by using these once daily regimens. However, no head-to-head trials comparing the safety and efficacy of fosamprenavir and atazanavir have been published. This prospective, randomized, open label 2-arm study will compare these two protease inhibitors for therapy of antiretroviral treatment-naïve HIV-infected patients. Patients who are successfully screened for eligibility will be randomized to receive tenofovir and emtricitabine plus either atazanavir (300mg qd) and ritonavir (100mg qd) or fosamprenavir (1400mg qd) and ritonavir (200mg qd). Participants will undergo assessment on day 1 and attend study visits at weeks 6, 12 and every 3 months until the completion of the study on week 96. "Antiretroviral Medication Self-Report" and "3-Day HIV Medication Self-Report" questionnaires will be applied at weeks 6, 12 and every 3 month, thereafter, until week 96. "Changes in Body Appearance" questionnaire will be applied at baseline and weeks 24, 48, 72, and 96.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Patient agrees to participate in the study by giving written informed consent.
* Documentation of HIV infection.
* No prior treatment with any anti-retroviral agent.
* CD4 cell count < 350 cells x mm3 or with an AIDS defining condition.
* Viral load > 1,000 copies/mL

Exclusion Criteria:

* Less than 18 years old.
* Current pregnancy or breastfeeding.
* Any previous antiretroviral regimen.
* Severe hepatic impairment that precludes the use of either study drug. This will be defined as any laboratory value of Grade 3 or 4 on the ACTG scale.
* Use of any contra-indicated medication as defined in the package insert for each drug.
* Any condition that, in the judgment of the investigator, precludes successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2004-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto C Arduino, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Thomas Street Health Center, Houston, Texas, United States

REFERENCES:
- [Background] Murphy RL, Sanne I, Cahn P, Phanuphak P, Percival L, Kelleher T, Giordano M. Dose-ranging, randomized, clinical trial of atazanavir with lamivudine and stavudine in antiretroviral-naive subjects: 48-week results. AIDS. 2003 Dec 5;17(18):2603-14. doi: 10.1097/00002030-200312050-00007. PMID 14685054
- [Background] Sax PE. Meeting notes from the 2nd International AIDS Society Conference on HIV Pathogenesis and Treatment. Atazanavir in treatment-experienced patients. AIDS Clin Care. 2003 Sep;15(9):78. PMID 14666914
- [Background] Bayes M, Rabasseda X, Prous JR. Gateways to clinical trials. Methods Find Exp Clin Pharmacol. 2003 Jul-Aug;25(6):483-506. PMID 12949633
- [Background] Goldsmith DR, Perry CM. Atazanavir. Drugs. 2003;63(16):1679-93; discussion 1694-5. doi: 10.2165/00003495-200363160-00003. PMID 12904086
- [Background] Rodriguez-French A, Boghossian J, Gray GE, Nadler JP, Quinones AR, Sepulveda GE, Millard JM, Wannamaker PG. The NEAT study: a 48-week open-label study to compare the antiviral efficacy and safety of GW433908 versus nelfinavir in antiretroviral therapy-naive HIV-1-infected patients. J Acquir Immune Defic Syndr. 2004 Jan 1;35(1):22-32. doi: 10.1097/00126334-200401010-00003. PMID 14707788
- [Background] SOLO trial results released. AIDS Patient Care STDS. 2003 Feb;17(2):95. doi: 10.1089/108729103321150827. No abstract available. PMID 12639292
- [Background] Falcoz C, Jenkins JM, Bye C, Hardman TC, Kenney KB, Studenberg S, Fuder H, Prince WT. Pharmacokinetics of GW433908, a prodrug of amprenavir, in healthy male volunteers. J Clin Pharmacol. 2002 Aug;42(8):887-98. doi: 10.1177/009127002401102803. PMID 12162471
- [Background] Vierling P, Greiner J. Prodrugs of HIV protease inhibitors. Curr Pharm Des. 2003;9(22):1755-70. doi: 10.2174/1381612033454441. PMID 12871195
- [Background] Mannheimer SB, Matts J, Telzak E, Chesney M, Child C, Wu AW, Friedland G; Terry Beirn Community Programs for Clinical Research on AIDS. Quality of life in HIV-infected individuals receiving antiretroviral therapy is related to adherence. AIDS Care. 2005 Jan;17(1):10-22. doi: 10.1080/09540120412331305098. PMID 15832830
- [Result] Holmes A, Lucke J, Maghidman S, Fernandez-Bussy S, Barnett B, Arduino R. Tenofovir associated nephrotoxicity is dose-dependent ritonavir administration a co-factor? XVI International AIDS Conference. Toronto, Canada. August 13-18, 2006. Abstract TUPE0085.
- [Result] Bell TK, Holmes A, McCormack OE, Barnett BJ, Arduino RC. Changing Genotypic Resistance Patterns and Demographics of Antiretroviral-Naïve HIV Patients in Houston: 1999-2006. 44th Annual Meeting of the Infectious Diseases Society of America (IDSA). Toronto, Canada. October 12-15, 2006. Abstract 975.
- [Result] Holmes A, Bell T, Barnett B, Arduino R. Emerging resistance mutations in once-daily ritonavir-boosted protease inhibitor-containing antiretroviral regimens. 44th Annual Meeting of the Infectious Diseases Society of America (IDSA). Toronto, Canada. October 12-15, 2006. Abstract 973.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled at a county clinic
Groups:
- Atazanavir: Atazanavir/ritonavir (300mg/100mg) once daily
- Fosamprenavir: Fosamprenavir/ritonavir (1400mg/100mg) once daily
Period: Overall Study
Arm/Group | Atazanavir | Fosamprenavir
Started | 39 | 37
Completed | 21 | 15
Not Completed | 18 | 22
Not completed — Lost to Follow-up | 12 | 17
Not completed — Death | 4 | 2
Not completed — Lack of Efficacy | 1 | 2
Not completed — no medicaiton dispensed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atazanavir | Fosamprenavir | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 33 | 71
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (9.7) | 48 (10) | 48 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 28 | 28 | 56
Region of Enrollment [Number; unit: participants]
  United States | 39 | 37 | 76

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patient With Viral Load Less Than 400 Copies/mL
Time Frame: 24 weeks
Measure: Number; unit: percentage
Arm/Group | Atazanavir | Fosamprenavir
Number analyzed (Participants) | 18 | 15
percentage | 89 | 73

2. Secondary Outcome: CD4 Cell Count Change From Baseline During Treatment.
Time Frame: 24 weeks.
Measure: Mean (Standard Deviation); unit: cell/mm3
Arm/Group | Atazanavir | Fosamprenavir
Number analyzed (Participants) | 18 | 15
cell/mm3 | 139 (119) | 117 (99)

ADVERSE EVENTS:
Arm/Group | Atazanavir | Fosamprenavir
Serious Adverse Events (participants affected / at risk) | 9/39 | 6/37
Other Adverse Events (participants affected / at risk) | 9/39 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Atazanavir (N=39) | Fosamprenavir (N=37)
Left perineal abscess (Gastrointestinal disorders) | 1 (1) | 0/0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
death (General disorders) | 3 (3) | 2 (2)
Steven's Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cryptococal meningitis (Infections and infestations) | 0 (0) | 1 (1)
Rupture hemorrhagic cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Seizure Disorder (Nervous system disorders) | 1 (5) | 0 (0)
Intracraneal Hypertension (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atazanavir (N=39) | Fosamprenavir (N=37)
hyperbilirrubinemia (Gastrointestinal disorders) | 7 (7) | 0 (0)
Increased LFTs (Hepatobiliary disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
High porportion of subject did not complete the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No